CLINICAL TRIAL: NCT01493115
Title: A Randomized, Double-blind, 3-sequence, 3-period Cross-over, Single-dose Study of a New Formulation of Insulin Glargine Compared to the Marketed Lantus® in Japanese Patients With Type 1 Diabetes Mellitus Using the Euglycemic Clamp Technique
Brief Title: Single Dose Study With a New Insulin Glargine Formulation and Lantus® in Japanese Patients With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PKD12270; U1111-1120-0463 (Other: UTN)
Record Dates: First submitted 2011-11-29; First posted 2011-12-15 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sequence 1 (Experimental): Reference (insulin glargine) - Test1 (insulin glargine - new formulation dose 1) - Test2 (insulin glargine - new formulation dose 2)
  Interventions: Drug: Insulin glargine HOE901; Drug: Insulin glargine - New formulation HOE901
- Sequence 2 (Experimental): Test1 (insulin glargine - new formulation dose 1) - Test2 (insulin glargine - new formulation dose 2) - Reference (insulin glargine)
  Interventions: Drug: Insulin glargine HOE901; Drug: Insulin glargine - New formulation HOE901
- Sequence 3 (Experimental): Test2 (insulin glargine - new formulation dose 2) - Reference (insulin glargine) - Test1 (insulin glargine - new formulation dose 1)
  Interventions: Drug: Insulin glargine HOE901; Drug: Insulin glargine - New formulation HOE901

INTERVENTIONS:
Drug: Insulin glargine HOE901 — Pharmaceutical form:solution for injection Route of administration: subcutaneous
  Other Names: Lantus®
Drug: Insulin glargine - New formulation HOE901 — Pharmaceutical form:solution for injection Route of administration: subcutaneous

SUMMARY:
Primary Objective:

To compare the pharmacodynamic properties of two different doses of a new insulin glargine formulation with 0.4 U/kg Lantus®

Secondary Objective:

To compare the pharmacokinetic properties of two different doses of a new insulin glargine formulation with 0.4 U/kg Lantus® To assess the safety and tolerability of a new insulin glargine formulation

DETAILED DESCRIPTION:
The study duration per patient will be 4 to 12 weeks including 3 treatment periods each separated by a wash-out period of 6-20 days

ELIGIBILITY:
Inclusion criteria:

* Japanese male or female subjects, between 20 and 65 years of age, inclusive, with type 1 diabetes mellitus for more than one year, as defined by the Japanese Diabetes Society
* Body weight between 50.0 kg and 95.0 kg
* Body Mass Index between 18.0 and 30.0 kg/m2 inclusive
* Stable insulin regimen for at least 2 months prior to study
* Certified as otherwise healthy for type 1 diabetes mellitus patient by assessment of medical history and physical examination
* Women of childbearing potential must have a negative pregnancy test and must use a highly effective method of birth control. During the entire study female subjects of child bearing potential must use two independent methods of contraception. The accepted double contraception methods include use of an intra-uterine device or hormonal contraception in addition to one of the following contraceptive options: 1) condom; 2) diaphragm 3) spermicide.

Exclusion criteria:

* Any history or presence of clinically relevant cardiovascular, pulmonary, gastro-intestinal, hepatic, renal, metabolic (apart from diabetes mellitus type 1), hematological, neurological, psychiatric, systemic (affecting the body as a whole), ocular, gynecologic (if female), or infectious disease; any acute infectious disease or signs of acute illness
* More than one episode of severe hypoglycemia with seizure, coma or requiring assistance of another person during the past 6 months
* Presence or history of a drug allergy or clinically significant allergic disease according to the Investigator's judgment
* Participation in a trial with any investigational drug during the past 4 months
* Symptoms of a clinically significant illness in the 3 months before the study, which, according to the investigator's opinion, could interfere with the purposes of the study
* Regular use of any medication other than insulins in the last month before study start with the exception of thyroid hormones, lipid-lowering and antihypertensive drugs, and, if female, with the exception of hormonal contraception or menopausal hormone replacement therapy; any vaccination within the last 28 days
* Known hypersensitivity to insulin glargine or excipients of the study drug
* Any history or presence of deep leg vein thrombosis or a frequent appearance of deep leg vein thrombosis in first degree relatives (parents, siblings or children)

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2011-11; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Glucose infusion rate | up to day 2 of each period

SECONDARY OUTCOMES:
Pharmacokinetic parameter : Cmax | up to day 2 of each period
Pharmacokinetic parameter : Tmax | up to day 2 of each period
Pharmacokinetic parameter : AUC | up to day 2 of each period
Number of patients with adverse events | up to day 3 of each period
Safety-related parameters including electrocardiogram, vital signs and laboratory tests | up to day 3 of each period

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site Number 392001, Fukuoka, Japan